CLINICAL TRIAL: NCT00212030
Title: Japan-Working Groups of Acute Myocardial Infarction for the Reduction of Necrotic Damage by a K-ATP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSSCJ-2; UMIN_ID:C000000089
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Data mining; Nicorandil; Randomized clinical trial; SNPs
MeSH Terms: interventions — Nicorandil

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: nicorandil
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nicorandil — (0∙067 mg/kg as a bolus, followed by 1∙67 μg/kg per min as a 24-h continuous intravenous infusion
  Arms: 1
Drug: placebo — Control
  Arms: 2

SUMMARY:
To evaluate whether nicorandil as an adjunctive therapy for AMI reduces myocardial infarct size and improves regional wall motion

DETAILED DESCRIPTION:
The benefits of percutaneous coronary intervention (PCI) in acute myocardial infarction (AMI) are limited by reperfusion injury. In animal models, nicorandil, a hybrid of an ATP-sensitive K+ (KATP) channel opener and nitrates, reduces infarct size, so the Japan-Working groups of acute myocardial Infarction for the reduction of Necrotic Damage by a K-ATP channel opener (J-WIND-KATP) designed a prospective, randomized, multicenter study to evaluate whether nicorandil reduces myocardial infarct size and improves regional wall motion when used as an adjunctive therapy for AMI.

Twenty-six hospitals in Japan are participating in the J-WIND-KATP study. Patients with AMI who are candidates for PCI are randomly allocated to receive either intravenous nicorandil or placebo. The primary end-points are (1) estimated infarct size and (2) left ventricular function. Single nucleotide polymorphisms (SNPs) that may be associated with the function of KATP-channel and the susceptibility of AMI to the drug will be examined. Furthermore, a data mining method will be used to design the optimal combined therapy for post-myocardial infarction (MI) patients.

It is intended that J-WIND-KATP will provide important data on the effects of nicorandil as an adjunct to PCI for AMI and that the SNPs information that will open the field of tailor-made therapy. The optimal therapeutic drug combination will also be determined for post-MI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-79 years
2. Chest pain of more than 30 min
3. 0.1 mV ST-segment elevation in 2 contiguous ECG leads
4. Admission to hospital within 12 h of symptom onset
5. First episode of AMI
6. Candidates for PCI

Exclusion Criteria:

1. History of old myocardial infarction
2. Left main coronary artery stenosis
3. Severe liver and/or kidney dysfunction
4. Suspected aortic dissection
5. History of coronary artery bypass graft
6. History of allergic response to drugs
7. Severe hypovolemia
8. Right ventricular infarction

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2001-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
estimated infarct size | 72hrs
left ventricular function (left ventricular ejection fraction and end-diastolic volume) and regional wall motion | 2-8weeks and 6-12months

SECONDARY OUTCOMES:
survival rate | 2.7years (median follow-up)
cardiovascular events (ie, cardiac death, nonfatal re-infarction, re-hospitalization because of cardiac disease, revascularization) | 2.7years (median follow-up)
reperfusion injury (ie, malignant ventricular arrhythmia during reperfusion periods, re-elevation of ST-segment, worsening of chest pain) | 24hrs
the association of SNPs of ANP-related genes with response to ANP treatment | 2.7years (median follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Masafumi Kitakaze, MD, PhD, Study Chair — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- National Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Background] Minamino T, Jiyoong K, Asakura M, Shintani Y, Asanuma H, Kitakaze M; J-WIND Investigators. Rationale and design of a large-scale trial using nicorandil as an adjunct to percutaneous coronary intervention for ST-segment elevation acute myocardial infarction: Japan-Working groups of acute myocardial infarction for the reduction of Necrotic Damage by a K-ATP channel opener (J-WIND-KATP). Circ J. 2004 Feb;68(2):101-6. doi: 10.1253/circj.68.101. PMID 14745142